CLINICAL TRIAL: NCT05100862
Title: A Phase 3 Randomized, Open-Label Multicenter Study of Zanubrutinib (BGB-3111) Plus Anti-CD20 Antibodies Versus Lenalidomide Plus Rituximab in Patients With Relapsed/Refractory Follicular or Marginal Zone Lymphoma
Brief Title: A Study of Zanubrutinib Plus Anti-CD20 Versus Lenalidomide Plus Rituximab in Participants With Relapsed/Refractory Follicular or Marginal Zone Lymphoma
Acronym: MAHOGANY
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3111-308; CTR20232545 (Registry Identifier: ChinaDrugTrials); 2022-502548-12-00 (Registry Identifier: EU CTIS)
Record Dates: First submitted 2021-09-27; First posted 2021-10-29 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Relapsed/Refractory Follicular Lymphoma; Marginal Zone Lymphoma
Keywords: Zanubrutinib; BGB-3111; Rituximab; Lenalidomide; Obinutuzumab
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone | interventions — zanubrutinib; Rituximab; Lenalidomide; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Follicular Lymphoma Arm A: Zanubrutinib plus Obinutuzumab (Experimental): Participants will receive zanubrutinib and Obinutuzumab. Following the completion of the combination treatment, participants will continue receiving zanubrutinib monotherapy until confirmed disease progression, unacceptable toxicity, withdrawal of consent, or study termination, whichever occurs first.
  Interventions: Drug: Zanubrutinib; Drug: Obinutuzumab
- Follicular Lymphoma Arm B: Lenalidomide plus Rituximab (Active Comparator): Participants will receive lenalidomide and rituximab.
  Interventions: Drug: Rituximab; Drug: Lenalidomide
- Marginal Zone Lymphoma Arm C: Zanubrutinib plus Rituximab (Experimental): Participants will receive zanubrutinib and rituximab. Following the completion of the combination treatment, participants will continue receiving zanubrutinib monotherapy until confirmed disease progression, unacceptable toxicity, withdrawal of consent, or study termination, whichever occurs first.
  Interventions: Drug: Zanubrutinib; Drug: Rituximab
- Marginal Zone Lymphoma Arm D: Lenalidomide plus Rituximab (Active Comparator): Participants will receive lenalidomide and rituximab.
  Interventions: Drug: Rituximab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Zanubrutinib — Zanubrutinib will be administered orally as two 80-milligram (mg) capsules twice a day (160 mg twice a day) or four 80-mg capsules once a day (320 mg once a day) continuously in repeated 28-day cycles.
  Other Names: BGB-3111; Brukinsa
  Arms: Follicular Lymphoma Arm A: Zanubrutinib plus Obinutuzumab; Marginal Zone Lymphoma Arm C: Zanubrutinib plus Rituximab
Drug: Rituximab — Rituximab will be administered intravenously at a dose of 375 mg/meter squared on Days 1, 8, 15, and 22 of Cycle 1 and on Day 1 of Cycles 2 to 5. Each cycle is 28 days in length.
  Other Names: Rituxan; MabThera; Ruxience; Truxima
  Arms: Follicular Lymphoma Arm B: Lenalidomide plus Rituximab; Marginal Zone Lymphoma Arm C: Zanubrutinib plus Rituximab; Marginal Zone Lymphoma Arm D: Lenalidomide plus Rituximab
Drug: Lenalidomide — Lenalidomide will be administered orally as 20-mg capsules (10 mg if creatinine clearance ≥ 30 mL/min but < 60 mL/min) once a day on Days 1 to 21 of each 28-day cycle for a total of 12 cycles.
  Other Names: Revlimid
  Arms: Follicular Lymphoma Arm B: Lenalidomide plus Rituximab; Marginal Zone Lymphoma Arm D: Lenalidomide plus Rituximab
Drug: Obinutuzumab — Obinutuzumab will be administered at a dose of 1000 mg on Cycle 1 Days 1, 8, 15 and then on Cycles 2 to 6 Day 1.
  Arms: Follicular Lymphoma Arm A: Zanubrutinib plus Obinutuzumab

SUMMARY:
The purpose of the study is to compare the efficacy of zanubrutinib plus obinutuzumab versus lenalidomide plus rituximab (R^2) in participants with relapsed/refractory (R/R) follicular lymphoma (FL), as measured by progression-free survival as determined by an independent review committee in accordance with the 2014 modification of the International Working Group on non-Hodgkin lymphoma (NHL) Criteria based on n positron emission tomography and computed tomography (PET/CT), and to compare the efficacy of zanubrutinib plus rituximab versus R^2 in participants with R/R marginal zone lymphoma (MZL), as measured by progression free survival (PFS) assessed by IRC in accordance with CT-based Lugano 2014 Criteria.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed grade 1-3a FL or MZL
* Previously treated with ≥ 1 line of systemic therapy including anti-CD20 agent. Must have a documented failure to achieve at least partial response during the most recent systemic therapy or documented progressive disease after the most recent systemic therapy
* Need for systemic therapy for FL or MZL
* Measurable disease by computed tomography or magnetic resonance imaging
* Adequate bone marrow, liver and renal function

Key Exclusion Criteria:

* Transformation to aggressive lymphoma
* Requiring ongoing need for corticosteroid treatment
* Clinically significant cardiovascular disease
* Prior malignancy within the past 2 years
* Active fungal, bacterial, and/or viral infection that requires systemic therapy
* Prior treatment with lenalidomide or drug from same class, if without response (partial or complete) or short remission duration (< 24 months)

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival As Determined By A Blinded Independent Review Committee (BIRC) | Approximately 78 months

SECONDARY OUTCOMES:
Progression-free Survival As Determined By Investigator Assessment | Approximately 87 months
Duration Of Response As Determined By BIRC And By Investigator Assessment | Approximately 87 months
Overall Response Rate As Determined By BIRC And By Investigator Assessment | Approximately 87 months
Complete Response Rate As Determined By BIRC And By Investigator Assessment | Approximately 87 months
Time To Response As Determined By BIRC And By Investigator Assessment | Approximately 87 months
Time to Next Ant-Lymphoma Treatment | Approximately 87 months
Overall Survival | Approximately 87 months
Health-related Quality Of Life (HRQoL) Using EORTC QLQ-C30) | Approximately 87 months
  HRQ0L assessed by The European Organization For Research On Treatment Of Cancer Quality Of Life Questionnaire-core 30 (EORTC QLQ-C30) consists of 30 questions that are associated with 5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, pain, and nausea and vomiting), and 6 single symptom items ( dyspnoea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The scores range from 0 to 100 and higher score indicates better quality of life.
HRQoL Using European Quality of Life 5 Dimension 5 Level Questionnaire [EQ 5D 5L) | Approximately 87 months
  The EQ-5D-5L is comprised of a descriptive module and a visual analogue scale. The EQ-5D-5L descriptive module comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The visual analogue scale records the respondent's self-rated health on a 0 to 100 scale, with 100 labeled "the best health you can imagine" and 0 labeled "the worst health you can imagine. Higher scores indicate better quality of life.
HRQoL Using National Comprehensive Cancer Network/Functional Assessment of Cancer Therapy Lymphoma Symptom Index-18 [FLymSI 18) | Approximately 87 months
  The FLymSI-18 is comprised of 18 questions which cover 4 sub-scales: physical symptoms, emotional symptoms, side effects, and functional well-being. Scores are based on the 5-level Likert scale with 5 possible responses ranging from 0 'Not at all' to 4 'Very much' and is divided into a total score. Higher score indicates better quality of life.
Number of Participants Experiencing Adverse Events (AEs) | From first dose to 28 days after the last dose of zanubrutinib or lenalidomide, 90 days after the last dose of obinutuzumab or rituximab, or until the date of confirmed disease progression, whichever comes later (Approximately 87 months)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene; Study Director, Principal Investigator — BeiGene
Locations (258):
- United States (31):
  - Ucsf Fresno University of California San Francisco Fresno, Fresno, California
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - Los Angeles Cancer Network, Los Angeles, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - Sharp Healthcare Sharp Memorial Hospital, San Diego, California
  - Baptist Md Anderson Cancer Center, Jacksonville, Florida
  - Northwest Georgia Oncology Centers Marietta, Marietta, Georgia
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Mission Cancer and Blood, Waukee, Iowa
  - Cancer Center of Kansas, Wichita, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Christus Highland Cancer Treatment Center, Shreveport, Louisiana
  - University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - American Oncology Partners of Maryland Pa, Bethesda, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Corewell Health the Michigan Cancer Consortium, Grand Rapids, Michigan
  - Hattiesburg Hematology and Oncology Clinic, Hattiesburg, Mississippi
  - University of Missouri Hospital, Ellis Fischel Cancer Center, Columbia, Missouri
  - Oncology Hematology Associates, Springfield, Missouri
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Iyengar Hematology Oncology Medical Center Pa, Bayonne, New Jersey
  - New York Cancer and Blood Specialists, Shirley, New York
  - Clinical Research Alliance, Inc, Westbury, New York
  - Levine Cancer Institute Wake Forest, Charlotte, North Carolina
  - Cancer Care Associates of York, York, Pennsylvania
  - Prairie Lakes Healthcare System, Watertown, South Dakota
  - Texas Oncology Baylorcharles A Sammons Cancer Center, Dallas, Texas
  - Md Anderson Cancer Center, Houston, Texas
  - Northeast Texas Cancer and Research Institute, Tyler, Texas
  - University of Washington, Seattle, Washington
  - Northwest Medical Specialties, Tacoma, Washington
- Argentina (2):
  - Hospital Aleman, CABA
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma Buenos Aires
- Australia (18):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Orange Health Hospital, Orange, New South Wales
  - Port Macquarie Base Hospital, Port Macquarie, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Sunshine Coast Hospital and Health Service, Birtinya, Queensland
  - Townsville University Hospital, Douglas, Queensland
  - Genesiscare North Adelaide, North Adelaide, South Australia
  - Monash Health, Clayton, Victoria
  - Epworth Freemasons, East Melbourne, Victoria
  - St Vincents Hospital Melbourne, Fitzroy, Victoria
  - Austin Health, Heidelberg, Victoria
  - Cabrini Hospital Malvern, Malvern East, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - La Trobe Regional Hospital, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
  - Perth Blood Institute, West Perth, Western Australia
- Austria (5):
  - Medizinische Universitatsklinik Innsbruck, Innsbruck
  - Uk St Poelten, Sankt Pölten
  - Medical Univeristy Vienna, Vienna
  - Hanusch Krankenhaus, Vienna
  - Wiener Gesundheitsverbund Klinik Ottakring, Vienna
- Belgium (4):
  - Institut Jules Bordet, Anderlecht
  - Az Sint Jan Brugge, Bruges
  - Universitair Ziekenhuis Gent, Ghent
  - University Hospitals Leuven, Leuven
- Brazil (22):
  - Hospital de Amor Barretos, Barretos
  - Clinica de Oncologia Reichow, Blumenau
  - Unesp Faculdade de Medicina Da Universidade Estadual Paulista Campus Botucatu, Botucatu
  - Instituto Dor de Pesquisa E Ensino Distrito Federal, Brasília
  - Universidade de Campinas Centro de Hematologia E Hemoterapia, Campinas
  - Fundacao Universidade de Caxias Do Sul, Caxias do Sul
  - Centro Integrado de Oncologia de Curitiba Ss Cionc, Curitiba
  - Hospital Erasto Gaertner, Curitiba
  - Centro de Ensino E Pesquisa Em Oncologia de Santa Catarina (Cepen), Florianópolis
  - Complexo Hospitalar de Niteroi, Niterói
  - Centro Gaucho Integrado de Oncologia Hospital Mae de Deus, Porto Alegre
  - Instituto Dor de Pesquisa E Ensino Pernambuco, Recife
  - Instituto Dor de Pesquisa E Ensino, Recife
  - Hospital Das Clinicas Da Faculdade de Medicina de Ribeirao Preto Usp, Ribeirão Preto
  - Instituto Americas Ensino, Pesquisa E Inovacao, Rio de Janeiro
  - Hospital Sao Rafaelinstituto Dor de Pesquisa E Ensino, Salvador
  - Ensino E Terapia de Inovacao Clinica Amo Etica, Salvador
  - Hospital Nove de Julho Dasa, São Paulo
  - Instituto Dor de Pesquisa E Ensino Sao Paulo, São Paulo
  - Hcfmusp Servico de Hematologia, Hemoterapia E Terapia Celular, São Paulo
  - Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein, São Paulo
  - Hospital Santa Rita de Cassia Afecc, Vitória
- Bulgaria (4):
  - Umhat Svgeorgi Ead, Plovdiv
  - Acibadem City Clinic Tokuda Umhat Ead, Department of Medical Oncology, Sofia
  - University Multiprofile Hospital For Active Treatment Saint Ivan Rilski, Sofia
  - NHATHD, Sofia
- Canada (11):
  - British Columbia Cancer Agency the Vancouver Centre, Vancouver, British Columbia
  - Newfoundland and Labrador Health Services, St. John's, Newfoundland and Labrador
  - Queen Elizabeth Ii Health Sciences Centre, Halifax, Nova Scotia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ciusss Du Saguenay Lac St Jean, Chicoutimi, Quebec
  - Centre Integre de Sante Et de Services Sociaux de Chaudiere Appalaches, Lévis, Quebec
  - Ciusss de Lest de Lile de Montreal Hopital Maisonneuve Rosemont, Montreal, Quebec
  - Unite de Recherche Clinique Du Cisss Des Laurentides, SaintJerome, Quebec
  - Ciusss de Lestrie Chus, Sherbrooke, Quebec
  - Chu de Quebec Universite Laval, Hopital de Lenfant Jesus, Centre Integre de Cancerologie (Cic), Québec
- China (38):
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University(Tongzhou), Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The First Peoples Hospital of Foshan, Foshan, Guangdong
  - Sun Yat Sen University Cancer Center, Guangzhou, Guangdong
  - Huizhou Central Peoples Hospital, Huizhou, Guangdong
  - Meizhou People Hospital, Meizhou, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Anyang Tumor Hospital, Anyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Peoples Hospital of Changde City, Changde, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Wuxi Peoples Hospital, Wuxi, Jiangsu
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - Jiangxi Province Cancer Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University Branch Xianghu, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - Peoples Hospital of Rizhao, Rizhao, Shandong
  - The Second Affiliated Hospital of Shandong First Medical University, Taian, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Dongyang Peoples Hospital, Dongyang, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Hospital of Jiaxing, Jiaxing, Zhejiang
  - Jinhua Municipal Central Hospital, Jinhua, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
- Czechia (2):
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Fakultni Nemocnice Olomouc, Olomouc
- France (8):
  - Hopital Prive Dantony, Departement Dhemathologie, Antony
  - Centre Hospitalier Le Mans, Le Mans
  - Chu Montpellier Hopital Saint Eloi, Montpellier
  - Hopital Larchet Chu Nice, Nice
  - Institut Curie, Paris
  - Necker University Hospital, Paris
  - Icans Institut de Cancerologie Strasbourg Europe, Strasbourg
  - Chu Nancy Hopital Brabois, VandoeuvrelesNancy
- JSC VIAN, Kutaisi, Georgia
- Germany (2):
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Ulm, Ulm
- Greece (4):
  - University Hospital of Alexandroupolis, Alexandroupoli
  - Evaggelismos, Athens
  - General Hospital of Athens Alexandra, Athens
  - University Hospital of Patra, Pátrai
- Ireland (2):
  - St Jamess Hospital, Dublin
  - University Hospital Waterford, Waterford
- Israel (7):
  - Assuta Ashdod Medical Center, Ashdod
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah En Karem Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Assuta Medical Center, Tel Aviv
  - Sourasky Tel Aviv Medical Center, Tel Aviv
- Italy (10):
  - Cro Irccs Aviano, Aviano
  - Irccs Azienda Ospedaliero Universitaria Bologna, Bologna
  - Aou Careggi, Servizio Sanitario Toscana, Florence
  - Istituto Europeo Di Oncologia, Milan
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Aou Maggiore Della Carita, Novara
  - Azienda Ospedaliera Di Padova, Padua
  - Irccs Policlinico San Matteo, Universita Degli Studi Di Pavi, Pavia
  - Arcispedale S Maria Nuova Ausl Reggio Emilia Hematology Unit, Reggio Emilia
  - Aou Santa Maria Della Misericordia Di Udine, Udine
- Japan (20):
  - Aichi Cancer Center Hospital Clinical Oncology, Nagoya, Aichi-ken
  - Chiba Cancer Center, Chiba, Chiba
  - Matsuyama Red Cross Hospital, Matsuyama, Ehime
  - Hiroshima Red Cross Hospital and Atomic Bomb Survivors Hospital, Hiroshima, Hiroshima
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Aiiku Hospital, Sapporo, Hokkaido
  - Kagoshima University Hospital, Kagoshima, Kagoshima-ken
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - University Hospital, Kyoto Prefectural Univ of Medicine, KyotoShi, Kyoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Kurashiki Central Hospital, Kurashikishi, Okayama-ken
  - Kansai Medical University Hospital, Hirakata, Osaka
  - Kindai University Hospital, Sakai, Osaka
  - Tokyo Metropolitan Komagome Hospital, Bunkyoku, Tokyo
  - National Cancer Center Hospital, ChuoKu, Tokyo
  - Cancer Institute Hospital of Jfcr, Kotoku, Tokyo
  - Yamagata University Hospital, Yamagata, Yamagata
  - Kumamoto University Hospital, Kumamoto
  - National Hospital Organization Okayama Medical Center, Okayama
  - Yokohama Municipal Citizens Hospital, Yokohama
- Poland (9):
  - Szpital Uniwersytecki Nr Im Dr Jana Biziela, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne Klinika Hematologii I Transplantologii, Gdansk
  - Pratia Onkologia Katowice, Katowice
  - Pratia McM Krakow, Krakow
  - Uniwersytecki Szpital Kliniczny W Poznaniu Oddzial Hematologii I Transplantacji Szpiku, Poznan
  - Wojewodzki Szpital Zespolony Im L Rydygiera W Toruniu, Torun
  - Centralny Szpital Kliniczny Uck Wum, Warsaw
  - Instytut Hematologii I Transfuzjologii, Warsaw
  - Narodowy Instytut Onkologii Im Marii Sklodowskiej Curie Hematology Unit, Warsaw
- Portugal (3):
  - Hospital de Braga, Braga
  - Instituto Portugues de Oncologia Do Porto Francisco Gentil, Epe, Porto
  - Unidade Local de Saude Gaia E Espinho, VILA NOVA de GAIA Porto
- Auxilio Mutuo Cancer Center, San Juan, Puerto Rico
- Romania (4):
  - Coltea Clinical Hospital, Bucharest
  - Institutul Oncologic Prof Dr Ion Chiricuta Cluj Napoca, ClujNapoca
  - Institutul Regional de Oncologie Iasi, Iași
  - Spitalul Clinic Judetean de Urgenta Bihor, Oradea
- South Africa (2):
  - Haemalife, Kuils River
  - Alberts Cellular Therapy, Pretoria
- South Korea (13):
  - Inje University Busan Paik Hospital, BusanjinGu, Busan Gwang'yeogsi
  - Dong A University Hospital, Seogu, Busan Gwang'yeogsi
  - Pusan National University Hospital, Seogu, Busan Gwang'yeogsi
  - Seoul National University Bundang Hospital, BundangGu SeongnamSi, Gyeonggi-do
  - Kyungpook National University Chilgok Hospital, BukGu, Gyeongsangbukdo
  - Gyeongsang National University Hospital, Jinju, Gyeongsangnam-do
  - Chonnam National University Hwasun Hospital, HwasunGun, Jeollanam-do
  - Samsung Medical Center, GangnamGu, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St Marys Hospital, SeochoGu, Seoul Teugbyeolsi
  - Severance Hospital Yonsei University Health System, SeodaemunGu, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center, SongpaGu, Seoul Teugbyeolsi
  - Soon Chun Hyang University Hospital Seoul, YongsanGu, Seoul Teugbyeolsi
- Spain (17):
  - Ico Badalona, Badalona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario Puerta Del Mar, Cadiz
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Institut Catala Doncologia Hospital Duran I Reynals, L'Hospitalet de Llobregat
  - Complejo Asistencial Universitario de Leon, León
  - Hospital de La Princesa, Madrid
  - Clinica Universidad de Navarra, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - H Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Clinico Universitario Virgen de La Arrixaca, Murcia
  - Clinica Universidad de Navarra Pamplona, Pamplona
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitari Mutua Terrassa, Terrassa
- Switzerland (4):
  - St Claraspital, Basel
  - Hfr Fribourg, Fribourg
  - Reseau Hospitalier Neuchatelois, La ChauxdeFonds
  - Universitatsspital Zurich, Zurich
- Turkey (Türkiye) (5):
  - Ankara University Medical Faculty, Ankara
  - Gazi University Medical School, AOCiftlii
  - Bagcilar Medipol Mega Hospital, Istanbul
  - Kocaeli Universitesi Tip Fakultesi, Kocaeli
  - Vkv American Hospital, Tevikiye
- United Kingdom (9):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - The Christie Hospital, Greater Manchester
  - Huddersfield Royal Infirmary, Huddersfield
  - Nhs Highland, Inverness
  - The Leeds Teaching Hospitals Nhs Trust, Leeds
  - Barts Health Nhs Trust, London
  - University College Hospital, London
  - Derriford Hospital, Plymouth
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/